CLINICAL TRIAL: NCT00986804
Title: Maintenance Therapy With Decitabine After Allogeneic Stem Cell Transplantation for Acute Myelogenous Leukemia and High-Risk Myelodysplastic Syndrome
Brief Title: Decitabine Maintenance for Acute Myelogenous Leukemia (AML) and Myelodysplastic Syndrome (MDS) Post Transplant
Acronym: AML MDS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-1126 / 201108378
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Leukemia, Myeloid, Acute; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Level 1 (Experimental): Decitabine 5.0 mg/m2/day on Days 1 thru 5 every 6 weeks for as many as 8 cycles.
  Interventions: Drug: Decitabine
- Level 2 (Experimental): Decitabine 7.5 mg/m2/day on Days 1 thru 5 every 6 weeks for as many as 8 cycles.
  Interventions: Drug: Decitabine
- Level 3 (Experimental): Decitabine 10.0 mg/m2/day on Days 1 thru 5 every 6 weeks for as many as 8 cycles.
  Interventions: Drug: Decitabine
- Level 4 (Experimental): Decitabine 15.0 mg/m2/day on Days 1 thru 5 every 6 weeks for as many as 8 cycles.
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine
  Other Names: Dacogen

SUMMARY:
Primary:

To determine the maximum tolerated dose and schedule of decitabine when administered as maintenance therapy after allogeneic hematopoietic stem cell transplantation (alloHSCT) performed for AML or high-risk MDS.

DETAILED DESCRIPTION:
Secondary:

* To determine the safety and tolerability of decitabine as maintenance therapy after alloHSCT.
* To determine the rates disease relapse, 1-year disease-free survival, and overall survival.
* To assess lymphoid and myeloid chimerism while on decitabine maintenance.
* To determine the incidence of acute and chronic GVHD.
* To assess immunologic reconstitution after alloHSCT.
* To assess changes in gene expression and methylation patterns following decitabine treatment
* To assess the effects of decitabine on immune reconstitution post transplant.
* To access the frequency of FoxP3+ CD3+/CD4+ and CD3+/CD8+ lymphocytes before and after decitabine treatment.

ELIGIBILITY:
Patient Screening Criteria and Enrollment Process

This is a single institution study at Washington University School of Medicine in St. Louis. Study population are patients >=18 years of age, with histologically confirmed AML or MDS according to World Health Organization (WHO) criteria undergoing alloHCST. All screening procedures are part the patients clinical care.

* Patients, or their legal authorized representative, will provide written informed consent for the study prior to alloHSCT, or through 100 days following alloHSCT
* Patients will undergo alloHSCT as per institutional guidelines. AlloHSCT may be performed using both related and unrelated donors, myeloablative or non-myeloablative preparative regimens, and with either peripheral blood or bone marrow as a source of graft.
* Patients who fulfill both the Inclusion Criteria and Exclusion Criteria in the period of ≥ 50 and ≤ 100 days after alloHSCT will be registered on the study and will receive decitabine maintenance. Bone marrow biopsy will be performed ≤ 14 days prior to starting decitabine to confirm remission. Any GVHD prophylaxis or therapy is allowed during the study.
* Patients who do not fulfill Inclusion Criteria are not eligible to be registered on the study and are considered screening failures.
* Study will include maximum of 32 evaluable patients.

Inclusion Criteria

* History of AML or MDS using WHO classification.
* >50 and <100 days following HLA-matched related or unrelated donor alloHSCT. Donors may be mismatched at single antigen at HLA-A, -B or -DR locus plus possible single antigen mismatch at HLA-C according to institution guidelines. Two-antigen mismatch at a single locus is not allowed.
* Age >=18 years.
* Bone marrow biopsy confirming complete remission after alloHSCT

  o Complete remission: less than 5% blasts in an aspirate bone marrow sample with a count of at least 200 nucleated cells, no blasts with Auer rods or persistence of extramedullary disease PLUS absolute neutrophil count (ANC) > 1,500/μL, platelet count ≥ 50,000/μL and no leukemic blasts in the peripheral blood.
* Platelet count ≥ 50,000/µL without platelet transfusion for 7 days and ANC ≥ 1,500/µL without colony stimulating factor support.
* Performance status < ECOG 2.
* Acceptable organ function defined as:

  * creatinine < 1.5 times the institutional ULN or creatinine clearance (calculated by the Cockroft and Gault method) ≥ 30 mL/min
  * bilirubin < 1.5 times the institutional ULN
  * AST, ALT and alkaline phosphatase < 2.5 times the institutional ULN.
* Each Patient or their legal authorized representative must sign an institutional review board/ethics committee-approved informed consent indicating their awareness of the investigational nature of this study.
* Female Subjects:
* Female of childbearing potential (FCBP*) must agree to use a reliable form of contraception or to practice complete abstinence from heterosexual intercourse for at least 28 days before starting study drug, while participating in the study, and for at least 28 days after discontinuation from the study. The methods of reliable contraception include intrauterine device (IUD), hormonal (birth control pills, injections, or implants), tubal ligation, partner's vasectomy, latex condom, diaphragm and cervical cap.
* FCBP must agree to pregnancy testing.
* FCBP must a negative pregnancy test prior to starting study drug.
* FCBP must agree to abstain from donating blood and/or egg during study participation and for at least 28 days after discontinuation from the study

  * A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., who has had menses at any time in the preceding 24 consecutive months).
* Male Subjects:
* Must agree to use a latex condom during sexual contact with FCBP while participating in the study and for at least 28 days following discontinuation from the study even if he has undergone a successful vasectomy
* Must agree to abstain from donating blood, semen, or sperm during study participation and for at least 28 days after discontinuation from the study.
* Must agree that if a pregnancy or a positive pregnancy test does occur in a female partner of a male study subject during study participation, study drug must be immediately discontinued and must immediately notify the principal investigator.

Exclusion Criteria

* History of previous alloHSCT prior to the current alloHSCT.
* Persistent AML or MDS after alloHSCT.
* Grade 3- 4 acute GVHD, See Appendix A.
* Positive serology for HIV.
* Pregnancy or nursing.
* Other cancers less than or equal to 2 years prior study entry except: basal cell carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the breast, prostate cancer stage T1a or T1b.
* Uncontrolled active infections requiring intravenous antibiotics.
* Clinically significant systemic illness (e.g. serious active infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), which, in the judgment of the Principal or Associate Investigator would compromise the patient's ability to tolerate protocol therapy.
* Known or suspected hypersensitivity to decitabine.
* Patients may not be receiving any other investigational agents.
* General or specific changes in patient's condition that render the patient unacceptable for further treatment in judgment of the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-12; Primary Completion 2014-05 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose and schedule of decitabine when administered as maintenance therapy after alloHSCT performed for AML or high-risk MDS. | Up to 6 weeks (completion of first cycle)

SECONDARY OUTCOMES:
To determine the safety and tolerability of decitabine as maintenance therapy after alloHSCT. | Up to 30 days after end of study (approximately 46 weeks)
To determine the rates disease relapse | Every 3 months for 2 years then every 6 months for 3 years
To assess lymphoid and myeloid chimerism while on decitabine maintenance. | End of cycle 3 (18 weeks)
To determine the incidence of acute GVHD. | End of study (42 weeks)
To assess immunologic reconstitution after alloHSCT. | End of study (42 weeks)
To assess changes in gene expression and methylation patterns following decitabine treatment | End of study (42 weeks)
To assess the effects of decitabine on immune reconstitution post transplant. | End of study (42 weeks)
To access the frequency of FoxP3+ CD3+/CD4+ and CD3+/CD8+ lymphocytes before and after decitabine treatment. | End of cycle 3 (18 weeks)
To determine the 1-year disease-free survival | 1 year
To determine overall survival. | Every 3 months for 2 years then every 6 months for 3 years
To determine the incidence of chronic GVHD. | End of study (42 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Iskra Pusic, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Blum W, Bruner-Klisovic R, Liu S, et al. Phase I Study of Low Dose Decitabine in Patients with Acute Myeloid Leukemia (AML): Pharmacokinetics (PK), Pharmacodynamics (PD), and Clinical Activity. ASH Annual Meeting Abstracts. 2005;106:1861-.
- [Background] Kantarjian H, Issa JP, Rosenfeld CS, Bennett JM, Albitar M, DiPersio J, Klimek V, Slack J, de Castro C, Ravandi F, Helmer R 3rd, Shen L, Nimer SD, Leavitt R, Raza A, Saba H. Decitabine improves patient outcomes in myelodysplastic syndromes: results of a phase III randomized study. Cancer. 2006 Apr 15;106(8):1794-803. doi: 10.1002/cncr.21792. PMID 16532500
- [Background] Choi J, Ritchey J, DiPersio J. Generation of Treg-Like Cells from CD4+CD25- T Cells Via Epigenetic Modification Using a Demethylating Agent Decitabine. ASH Annual Meeting Abstracts. 2007;110:62-.
- [Background] De Lima M, de Padua Silva L, Giralt S, et al. Maintenance Therapy with Low-Dose Azacitidine (AZA) after Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) for Relapsed or Refractory AML or MDS: A Dose and Schedule Finding Study. ASH Annual Meeting Abstracts. 2008;112:1134-.
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu